CLINICAL TRIAL: NCT06000280
Title: Evaluation of Macular Thickness in Patients With Glaucoma in Use of Topical Prostaglandin Analogue Undergoing Trabeculectomy With Mitomycin C
Brief Title: Evaluation of Retina in Patients With Glaucoma Using Topical Prostaglandins Undergoing Trabeculectomy Surgery
Acronym: TRAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, David Leonardo Cruvinel Isaac, Clinical Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEROF
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma
Keywords: prostaglandin analogue; macular edema; trabeculectomy
MeSH Terms: conditions — Glaucoma; Macular Edema

STUDY DESIGN:
Intervention Model Description: This is a randomized, prospective and comparative clinical trial. Both the surgeon (the only one) and the technician responsible for the exams were blinded to the study groups. The patients (one or both eyes) included were from the glaucoma outpatient clinic of the Fundação Banco de Olhos de Goiás (FUBOG) or the Reference Center in Ophthalmology (CEROF) of the Federal University of Goiás (UFG) between the years 202 and 2022. All patients with glaucoma with indication for Trab with MMC and in clinical use of any PA eye drops (latanoprost, travoprost, bimatoprost or tafluprost) in the eye to be operated on for at least 6 months were considered for inclusion.
  The study adhered to the principles of the Declaration of Helsinki and was authorized by the Research Ethics Committee of the UFG, under the Certificate of Presentation for Ethical Appreciation NUMBER 40055620.8.1001.5083. All those included voluntarily agreed to participate by signing the Free and Informed Consent Form.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The techinician who performed the exams (Optical Coherence Tomography and Visual Field)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): The Study group refers to patients who are using topical prostaglandins analogues
  Interventions: Procedure: Trabeculectomy surgery
- Control group (Placebo Comparator): The Control group refers to patients who discontinued the use of topical prostaglandins analogues
  Interventions: Procedure: Trabeculectomy surgery

INTERVENTIONS:
Procedure: Trabeculectomy surgery — The Trabeculectomy aims to create a permanent drainage outflow channel for the aqueous humor, connecting the anterior chamber to the sub-Tenon's space, using mitomycin C consisted of opening the conjunctival base of the fornix and applying mitomycin C 0.4 mg/ml for 2 minutes. The trabeculectomy techniques require controlled outflow of aqueous humor through a sclerostomy and a partial-thickness scleral flap to form a subconjunctival bleb. The protected strength of the flap, with or without sutures, and the strength of the episcleral tissue determine the final IOP.

SUMMARY:
The aim of this study was to verify whether prostaglandin analogue (PA) eye drops influence the retinal thickness of glaucomatous patients undergoing trabeculectomy (TRAB) surgery. We selected eyes of patients with glaucoma with surgical indication for TRAB who were using PA eye drops and without previous retinal alterations, from the Centro de Referência em Oftalmologia (CEROF) from the Federal University of Goiás and Fundação Banco de Olhos de Goiás (FUBOG). Patients were divided into 2 groups: the study group (SG) and the control group (CG). In the CG, the PA was suspended between 30 and 60 days before the preoperative exams were performed (maximum of 15 days before surgery for both groups). All patients included were submitted to various eye exams before the procedure, and postoperatively on 3 occasions: 1 to 3 days ("PO1"), 6 to 9 days ("PO7") and 27 to 30 days ("PO30") after surgery.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to verify whether topical prostaglandin analogue (PA) influence the macular thickness of glaucomatous patients undergoing trabeculectomy (TRAB) with Mitomycin C (MMC) .

Design:This is a randomized, prospective, comparative clinical trial with a single surgeon and masked to the study group.

Methods: We prospectively selected 40 eyes of patients with glaucoma with surgical indication for TRAB with MMC (0.4 mg/ml for 2 min) who were using prostaglandin analogue (PA) eye drops and without previous macular alterations, from the Centro de Referência em Oftalmologia (CEROF) from the Federal University of Goiás and Fundação Banco de Olhos de Goiás (FUBOG). The research had as inclusion criteria: patients with at least 18 years of age with Primary Glaucoma (Primary Open Angle Glaucoma, Primary Closed Angle Glaucoma, Normal Pressure Glaucoma, Pigmentary Glaucoma, Pseudoesfoliative Glaucoma), with changes in the visual field, typical defect compatible with glaucomatous lesion and/or typical anatomical impairment of the optic disc or retinal nerve fiber layer (such as Hoyt's sign, optic disc cupping ratio greater than 0.7, localized defect in the neural rima, or cupping asymmetry), who had an indication for TRAB with MMC at the physician's discretion (target IOP not established with maximum tolerable clinical medication and/or impossibility of using medication due to allergies and/or financial conditions). To be included, the operated eyes needed a reduction in IOP of at least 20% in relation to the baseline IOP in the last postoperative period (PO 30), and absence of the use of any ocular hypotensive medication. Exclusion criteria were any pathology that could interfere with the test results, such as: cataracts, corneal edema (such as leucoma, ulcers, keratopathies); poor quality of the OCT scan (signal strength ≤ 5/10); any past macular pathology (such as macular hole, diabetic maculopathy, age-related macular disease); use of diamox; advanced glaucoma with maximal therapy; advanced glaucoma with impaired fixation; any surgical complications including hypotonia (IOP < 6 mmHg) at any assessment; performing combined cataract and glaucoma surgery; history of cataract surgery less than 6 months ago; need for surgical reintervention during follow-up for any reason; and need for reintroduction of topical antiglaucoma therapy during follow-up. Eligible volunteers were previously randomized through the website www.randomization.com into 2 groups: study group (SG) and control group (CG). The initial objective was to include 40 eyes, 20 per group.

In the SG, patients were instructed to keep using eyedrops (including PA) until the day of surgery. In the CG, patients were instructed to suspend the PA between 30-60 days after the preoperative exams were performed, which were performed a maximum of 15 days before surgery for both groups. In the CG, patients were instructed to use 01 drop of carmellose sodium 5mg/ml at the same time they used the AP before its suspension. Pseudophakic patients for more than six months were included in each group in the order of previous randomization. In the CG, patients were informed to keep the eye drops in use, and to add the other classes of ocular hypotensive drugs, if they were not using them (except miotics and oral acetazolamide), with the aim of at least remedying the loss of the ocular hypotensive effect of the PA. The individuals were evaluated, including best corrected visual acuity by the Snellen chart, slit lamp biomicroscopy (XCELL 255, Reichert Inc., Depew, NY, USA), intraocular pressure (IOP) measured in a calibrated Goldmann tonometer (CT210, Reichert Inc. , Depew, NY, USA), gonioscopy with a 4-mirror Goldman lens (Volk Optical Inc, Mentor, OH, USA), fundoscopy under mydriasis with a 78D lens (Volk Optical Inc, Mentor, OH, USA), indirect binocular ophthalmoscopy with 2.0D lens (Volk Optical Inc, Mentor, OH, USA) and Optical Coherence Tomography (OCT) with Cirrus 4000 (Zeiss Inc.), macular protocol (macular thickness and ganglion cell analysis) preoperatively ( maximum of 15 days before surgery), and postoperatively on 3 occasions: 1 to 3 days ("PO1"), 6 to 9 days ("PO7") and 27 to 30 days ("PO30"). All tests were performed by the same technician, who was trained and experienced to carry them out. All patients underwent visual field examinations (Humphrey Field, model HFA II ÿ750, Carl Zeiss-Meditec, Dublin, California, USA) prior to surgery with the Swedish Interactive Threshold Algorithm (SITA) Standard 24-2 strategy, at most up to 2 months before the procedure. Macular thickness was evaluated by spectral domain Optical Coherence Tomography (OCT) obtained using the Cirrus 4000 apparatus (Zeiss Inc.), macular scanning protocol (macular thickness and ganglion cell analysis). Calculations were made based on data from the Ganglion cell analytical program and Macular Thickness: Macular cube (6 x 6 mm - 512 A-scans x 128 B-scans centered on the fovea). The macular thickness map using the 1mm, 3mm, and 6mm circles from the Early Treatment Diabetic Retinopathy Study (ETDRS) was used to assess the thickness of the 9 subfields. The regions were designated as: parafoveal (subfields of the 3 mm rings) and perifoveal (subfields of the 6 mm rings) superior, inferior, temporal and nasal in addition to the central subfield. OCT images were excluded if the signal strength was ≤5/10, and a new scan was immediately performed. Trabeculectomy using mitomycin C consisted of opening the conjunctival base of the fornix and applying mitomycin C 0.4 mg/ml for 2 minutes, as previously described. The postoperative regimen in both groups included the use of 1% Prednisolone eye drops (Ster® União Química Farmacêutica Nacional S/A., Pouso Alegre, MG, Brazil) starting every 2 hours, with a weekly reduction for 6 weeks ( 4/4 h, followed by 6/6 h, then every 8 h, 12/12 h and once a day), Moxifloxacin eye drops (Vigamox®, AlconLabs, Fort Worth, TX, USA) every 6 h for 10 days.

Statistical analysis was performed using the Statistical Package for Social Sciences program (IBM Corporation, Armonk, USA) version 26.0. The characterization of the sample was performed using absolute frequency, relative frequency, mean, standard deviation, median, minimum and maximum. Student's t test and Pearson's chi-square test were applied to the distribution of profile and macular parameters in groups with and without prostaglandin. Data normality was verified using the Shapiro-Wilk test. The delta and percentage variation were calculated at PO1, PO7 and PO30 in relation to the preoperative period. Correlation analysis was performed between thickness deltas with visual field Mean Deviation (MD) and IOP in groups with and without prostaglandin, weighted the effect of lens classification (partial correlation). The significance level adopted was 5% (p < 0.05).

Initially, 40 eyes were randomly assigned to the study, of which 17 were excluded because they did not meet the eligibility criteria for the study postoperatively. Among these, 4 patients did not undergo OCT at PO1, 4 patients did not undergo OCT at PO7, 2 patients did not undergo OCT at PO30, 1 patient had a signal ≤ 5/10 of OCT at all visits, even with several repetitions of the examinations, 3 patients underwent surgical reintervention during follow-up (suture dehiscence), 2 patients had hypotonia, finally 1 patient did not present IOP reduction by at least 20% of baseline. Thus, as there was a significant reduction in the number of patients initially estimated for the sample, a new randomization was performed, using the same initial randomization process described above to achieve this objective. In the end, the evaluated sample consisted of 40 eyes from 37 patients, 20 eyes per group (20 eyes from 18 patients in the CG and 20 eyes from 19 patients in the SG).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnose's of Primary Glaucoma

  * Primary Open Angle Glaucoma
  * Primary Closed Angle Glaucoma
  * Normal Pressure Glaucoma
  * Pigmentary Glaucoma
  * Pseudosfoliative Glaucoma)
* Changes in the visual field
* Typical defect compatible with glaucomatous lesion and/or typical anatomical impairment of the optic disc or retinal nerve fiber layer

  * Hoyt's sign
  * Optic disc cupping ratio greater than 0.7
  * Defect located in the neural rim or cupping asymmetry
* Indication for TRAB with MMC at the physician's discretion (target IOP not established with maximum tolerable clinical medication or impossibility of using medication due to allergies and/or financial conditions)
* The operated eyes needed a reduction in IOP by at least 20% in relation to the baseline IOP in the last postoperative period (PO30)
* Absence of the use of any ocular hypotensive medication.

Exclusion Criteria:

* Any pathology that could interfere with the test results

  * cataract (crystalline opacity)
  * corneal edema (such as leucoma, ulcers, keratopathies)
  * poor quality of exams (≤ 5/10)
  * any past macular pathology (such as macular hole, diabetic maculopathy, age related macular disease);
* Use of diamox
* Advanced glaucoma with maximal therapy
* Advanced glaucoma with impaired fixation
* Any surgical complications including hypotonia (IOP < 6 mmHg) at any assessment
* Performing combined cataract and glaucoma surgery
* History of cataract surgery less than 6 months ago
* Need for surgical reintervention during follow-up for any reason
* Need for reintroduction of topical antiglaucoma therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals self-identified as male and female were eligible for the study.
Enrollment: 37 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Previous use of prostaglandins does not change macular thickness after trabeculectomy | Measurements were performed at preop (up to 15 days before the intervention), 1 to 3 days ("PO1"), 6 to 9 days ("PO7") and 27 to 30 days ("PO30") after surgery.
  The absolute variation of each variable of the macular parameters OCT in relation to the pre-op was performed and its comparison between the groups at different moments. There was equivalence in most of the evaluated comparisons. Considering the variation between pre-op and PO30, only the upper parafoveal thickness was statistically different between groups (p= 0.01). Taking into account the difference in percentage analyzing pre-op vs. PO30, only the superior parafoveal thickness showed statistical significance between groups (p=0.01).

SECONDARY OUTCOMES:
The presence of the lens did not influence the correlations | Measurements were performed at preop (up to 15 days before the intervention) and 27 to 30 days ("PO30") after surgery.
  Correlations were performed between the deltas of the thicknesses of the macular parameters between the preoperative period and the PO30 within the groups with the possible confounding factors (MD and IOP) and also controlling the intensity of the lens effect (partial correlation). There was no significant correlation in the other tests performed, as well as in relation to the possible influence of the crystalline lens in each of them.

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Magacho dos Santos Silva, Doctor, Study Director — Universidade Federal de Goias
Locations (1):
- Centro de Referencia em Oftalmologia, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data collected in the exams performed in the study and the data of the results will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be shared 6 months after publication
Access Criteria: Data sharing can be done after the consent of the main investigator of the study signed and sent by e-mail. Study principal investigator will review sharing requests
URL: https://www.gov.br/governodigital/pt-br/governanca-de-dados/regras-de-compartilhamento_v1-0.pdf

REFERENCES:
- [Background] Motero Carrasco J. [A comparative study of the efficacy of lisinopril versus quinapril in controlling light to moderate arterial hypertension. A follow-up with ABPM]. Rev Esp Cardiol. 1995 Nov;48(11):746-53. Spanish. PMID 8532944
- [Background] Yonekawa Y, Kim IK. Pseudophakic cystoid macular edema. Curr Opin Ophthalmol. 2012 Jan;23(1):26-32. doi: 10.1097/ICU.0b013e32834cd5f8. PMID 22134362
- [Background] Vessani R, Frota T, Shigetomi G, Correa P, Mariottoni EB, Tavares I. Structural Changes in the Optic Disc and Macula Detected by Swept-Source Optical Coherence Tomography After Surgical Intraocular Pressure Reduction in Patients with Open-Angle Glaucoma. Clin Ophthalmol. 2021 Jul 14;15:3017-3026. doi: 10.2147/OPTH.S317190. eCollection 2021. PMID 34285468
- [Background] Francoz M, Fenolland JR, Giraud JM, El Chehab H, Sendon D, May F, Renard JP. Reproducibility of macular ganglion cell-inner plexiform layer thickness measurement with cirrus HD-OCT in normal, hypertensive and glaucomatous eyes. Br J Ophthalmol. 2014 Mar;98(3):322-8. doi: 10.1136/bjophthalmol-2012-302242. Epub 2013 Dec 4. PMID 24307717
- [Background] Lavinsky F, Wu M, Schuman JS, Lucy KA, Liu M, Song Y, Fallon J, de Los Angeles Ramos Cadena M, Ishikawa H, Wollstein G. Can Macula and Optic Nerve Head Parameters Detect Glaucoma Progression in Eyes with Advanced Circumpapillary Retinal Nerve Fiber Layer Damage? Ophthalmology. 2018 Dec;125(12):1907-1912. doi: 10.1016/j.ophtha.2018.05.020. Epub 2018 Jun 19. PMID 29934267
- [Background] Klink T, Lieb WE, Gobel W. [Early and late findings with optical coherence tomography (OCT) in patients with postoperative hypotonia]. Ophthalmologe. 2000 May;97(5):353-8. doi: 10.1007/s003470050536. German. PMID 10892280
- [Background] Kim WJ, Kim KN, Sung JY, Kim JY, Kim CS. Relationship between preoperative high intraocular pressure and retinal nerve fibre layer thinning after glaucoma surgery. Sci Rep. 2019 Sep 25;9(1):13901. doi: 10.1038/s41598-019-50406-7. PMID 31554879
- [Background] Kadziauskiene A, Strelkauskaite E, Mockeviciute E, Asoklis R, Lesinskas E, Schmetterer L. Changes in macular thickness after trabeculectomy with or without adjunctive 5-fluorouracil. Acta Med Litu. 2017;24(2):93-100. doi: 10.6001/actamedica.v24i2.3489. PMID 28845126
- [Background] Raghu N, Pandav SS, Kaushik S, Ichhpujani P, Gupta A. Effect of trabeculectomy on RNFL thickness and optic disc parameters using optical coherence tomography. Eye (Lond). 2012 Aug;26(8):1131-7. doi: 10.1038/eye.2012.115. Epub 2012 Jun 22. PMID 22722487
- [Background] Silva D, Lopes AS, Henriques S, Lisboa M, Pinto S, Trancoso Vaz F, Prieto I. Changes in choroidal thickness following trabeculectomy and its correlation with the decline in intraocular pressure. Int Ophthalmol. 2019 May;39(5):1097-1104. doi: 10.1007/s10792-018-0918-y. Epub 2018 Apr 16. PMID 29663109
- [Background] Diaconita V, Quinn M, Jamal D, Dishan B, Malvankar-Mehta MS, Hutnik C. Washout Duration of Prostaglandin Analogues: A Systematic Review and Meta-analysis. J Ophthalmol. 2018 Sep 27;2018:3190684. doi: 10.1155/2018/3190684. eCollection 2018. PMID 30363694
- [Background] Mishima H, Masuda K, Miyake K. The putative role of prostaglandins in cystoid macular edema. Prog Clin Biol Res. 1989;312:251-64. No abstract available. PMID 2678143
- [Background] Taheri PA, Karamanoukian H, Gibbons K, Waldman N, Doerr RJ, Hoover EL. Can patients with minor head injuries be safely discharged home? Arch Surg. 1993 Mar;128(3):289-92. doi: 10.1001/archsurg.1993.01420150043008. PMID 8442684
- [Background] Gupta P, Sidhartha E, Tham YC, Chua DK, Liao J, Cheng CY, Aung T, Wong TY, Cheung CY. Determinants of macular thickness using spectral domain optical coherence tomography in healthy eyes: the Singapore Chinese Eye study. Invest Ophthalmol Vis Sci. 2013 Dec 5;54(13):7968-76. doi: 10.1167/iovs.13-12436. PMID 24222307
- [Background] Lichter PR. Variability of expert observers in evaluating the optic disc. Trans Am Ophthalmol Soc. 1976;74:532-72. PMID 867638
- [Background] Manabe K, Matsuoka Y, Tanito M. Incidence of macular edema development after filtration surgery. Graefes Arch Clin Exp Ophthalmol. 2020 Jun;258(6):1343-1345. doi: 10.1007/s00417-020-04624-9. Epub 2020 Feb 13. No abstract available. PMID 32055953
- [Background] Belyea DA, Dan JA, Lieberman MF, Stamper RL. Midterm follow-up results of combined phacoemulsification, lens implantation, and mitomycin-C trabeculectomy procedure. J Glaucoma. 1997 Apr;6(2):90-8. PMID 9098816
- [Background] Sesar A, Cavar I, Sesar AP, Geber MZ, Sesar I, Laus KN, Vatavuk Z, Mandic Z. Macular thickness after glaucoma filtration surgery. Coll Antropol. 2013 Sep;37(3):841-5. PMID 24308226
- [Background] Karasheva G, Goebel W, Klink T, Haigis W, Grehn F. Changes in macular thickness and depth of anterior chamber in patients after filtration surgery. Graefes Arch Clin Exp Ophthalmol. 2003 Mar;241(3):170-5. doi: 10.1007/s00417-003-0628-6. Epub 2003 Feb 20. PMID 12644938
- [Background] Pitale PM, Chatha U, Patel V, Gupta L, Waisbourd M, Pro MJ. Changes in macular thickness following glaucoma surgery. Int J Ophthalmol. 2016 Aug 18;9(8):1236-7. doi: 10.18240/ijo.2016.08.24. eCollection 2016. No abstract available. PMID 27588282
- [Background] Demirtas AA, Karahan M, Erdem S, Aslan Kaya A, Keklikci U. Long-term effects of trabeculectomy in primary open-angle glaucoma on segmented macular ganglion cell complex alterations. Int Ophthalmol. 2021 Jun;41(6):2249-2263. doi: 10.1007/s10792-021-01840-y. Epub 2021 Apr 21. PMID 33880684
- [Background] Nilforushan N, Loni S, Abdolalizadeh P, Miraftabi A, Banifatemi M, Rakhshan R, Jafari S, Abolfathzadeh N. Early Macular Thickness Changes after Trabeculectomy and Combined Phaco-Trabeculectomy. J Curr Ophthalmol. 2022 Jul 26;34(2):160-166. doi: 10.4103/joco.joco_333_21. eCollection 2022 Apr-Jun. PMID 36147280
- [Background] Wagner FM, Schuster AK, Kianusch K, Stingl J, Pfeiffer N, Hoffmann EM. Long-term success after trabeculectomy in open-angle glaucoma: results of a retrospective cohort study. BMJ Open. 2023 Feb 3;13(2):e068403. doi: 10.1136/bmjopen-2022-068403. PMID 36737088
- [Background] Koike KJ, Chang PT. Trabeculectomy: A Brief History and Review of Current Trends. Int Ophthalmol Clin. 2018 Summer;58(3):117-133. doi: 10.1097/IIO.0000000000000231. No abstract available. PMID 29870414
- [Background] Hollo G. The side effects of the prostaglandin analogues. Expert Opin Drug Saf. 2007 Jan;6(1):45-52. doi: 10.1517/14740338.6.1.45. PMID 17181451
- [Background] Alm A. Latanoprost in the treatment of glaucoma. Clin Ophthalmol. 2014 Sep 26;8:1967-85. doi: 10.2147/OPTH.S59162. eCollection 2014. PMID 25328381
- [Background] van der Valk R, Webers CA, Schouten JS, Zeegers MP, Hendrikse F, Prins MH. Intraocular pressure-lowering effects of all commonly used glaucoma drugs: a meta-analysis of randomized clinical trials. Ophthalmology. 2005 Jul;112(7):1177-85. doi: 10.1016/j.ophtha.2005.01.042. PMID 15921747
- [Background] Gazzard G, Konstantakopoulou E, Garway-Heath D, Garg A, Vickerstaff V, Hunter R, Ambler G, Bunce C, Wormald R, Nathwani N, Barton K, Rubin G, Buszewicz M; LiGHT Trial Study Group. Selective laser trabeculoplasty versus eye drops for first-line treatment of ocular hypertension and glaucoma (LiGHT): a multicentre randomised controlled trial. Lancet. 2019 Apr 13;393(10180):1505-1516. doi: 10.1016/S0140-6736(18)32213-X. Epub 2019 Mar 9. PMID 30862377
- [Background] Leske MC, Heijl A, Hyman L, Bengtsson B, Komaroff E. Factors for progression and glaucoma treatment: the Early Manifest Glaucoma Trial. Curr Opin Ophthalmol. 2004 Apr;15(2):102-6. doi: 10.1097/00055735-200404000-00008. PMID 15021220
- [Background] Prum BE Jr, Rosenberg LF, Gedde SJ, Mansberger SL, Stein JD, Moroi SE, Herndon LW Jr, Lim MC, Williams RD. Primary Open-Angle Glaucoma Preferred Practice Pattern((R)) Guidelines. Ophthalmology. 2016 Jan;123(1):P41-P111. doi: 10.1016/j.ophtha.2015.10.053. Epub 2015 Nov 12. PMID 26581556
- [Background] Weinreb RN, Aung T, Medeiros FA. The pathophysiology and treatment of glaucoma: a review. JAMA. 2014 May 14;311(18):1901-11. doi: 10.1001/jama.2014.3192. PMID 24825645
- [Background] Schuster AK, Wagner FM, Pfeiffer N, Hoffmann EM. Risk factors for open-angle glaucoma and recommendations for glaucoma screening. Ophthalmologe. 2021 Jul;118(Suppl 2):145-152. doi: 10.1007/s00347-021-01378-5. Epub 2021 Apr 21. PMID 33881589
- [Background] Flaxman SR, Bourne RRA, Resnikoff S, Ackland P, Braithwaite T, Cicinelli MV, Das A, Jonas JB, Keeffe J, Kempen JH, Leasher J, Limburg H, Naidoo K, Pesudovs K, Silvester A, Stevens GA, Tahhan N, Wong TY, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global causes of blindness and distance vision impairment 1990-2020: a systematic review and meta-analysis. Lancet Glob Health. 2017 Dec;5(12):e1221-e1234. doi: 10.1016/S2214-109X(17)30393-5. Epub 2017 Oct 11. PMID 29032195
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Causes of blindness and vision impairment in 2020 and trends over 30 years, and prevalence of avoidable blindness in relation to VISION 2020: the Right to Sight: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e144-e160. doi: 10.1016/S2214-109X(20)30489-7. Epub 2020 Dec 1. PMID 33275949
- See also: Centro de Referencia em Oftalmologia — https://cerof.ufg.br
- Available data/document: Informed Consent Form: Repositorio — http://repositorio.bc.ufg.br — Repositorio da Biblioteca Central da Universidade Federal de Goias